CLINICAL TRIAL: NCT02377193
Title: Prospective, Multicenter, Randomized, Evaluating Two Induction Therapies With Simulect® Versus ATG® Fresenius Associated With Tacrolimus and Myfortic® in the Prevention of Treatment Failure, in Sensitized Renal Transplant
Brief Title: Simulect Versus ATG in Sensitized Renal Transplant Patient
Acronym: SATIR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Neovii Biotech (Industry); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12 484 03
Record Dates: First submitted 2014-06-11; First posted 2015-03-03 (Estimated); Last update posted 2025-12-10 (Actual); Status verified 2017-10

CONDITIONS: Renal Transplant Rejection
Keywords: kidney transplant; luminex method; simulect ATG; immunosuppression
MeSH Terms: interventions — Basiliximab; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Simulect (Experimental): Simulect IV 40 mg D0 and D4
  Interventions: Drug: Simulect
- ATG Fresenius (Active Comparator): ATG IV min dose 3 mg/ kg/ day D0, D1, D3, D5
  Interventions: Drug: ATG Fresenius

INTERVENTIONS:
Drug: Simulect — Simulect IV 40 mg/day D0 and D4
  and oral use Tacrolimus 0.1 mg/ kg/ day + Myfortic 720 to 1440mg + Corticosteroids 5mg
  Other Names: Simulect IV 40 mg/day D0 and D4; and oral use Tacrolimus 0.1 mg/ kg/ day +; Myfortic 720 to 1440mg +; Corticosteroids 5mg
  Arms: Simulect
Drug: ATG Fresenius — Simulect IV 40 mg/day D0 and D4 and oral use Tacrolimus 0.1 mg/ kg/ day + Myfortic 720 to 1440mg + Corticosteroids 5mg
  Other Names: Simulect IV 40 mg/day D0 and D4; and oral use Tacrolimus 0.1 mg/ kg/ day +; Myfortic 720 to 1440mg +; Corticosteroids 5mg
  Arms: ATG Fresenius

SUMMARY:
Induction therapy by either T-cell depleting polyclonal antibodies such as anti-thymocyte globulins (ATG) or non-depleting anti-interleukine 2 receptor monoclonal antibodies (anti-CD25 moAb: basiliximab or daclizumab) are used to prevent acute rejection, especially in highly sensitized patients. Both induction therapy regimens have a different tolerance profile. Infections and haematological side-effects are more frequently reported in patients receiving ATG.

The aim of the pilot study is to evaluate ATG and basiliximab induction therapy in de novo sensitized kidney-transplant patients (incompatible grafts rate ≥ 50%) without donor specific antibodies (DSAs) detected by Luminex.

DETAILED DESCRIPTION:
Acute rejection after kidney transplantation can lead to graft loss by irreversible acute rejection or to interstitial fibrosis/ tubular atrophy that can induce graft loss. Induction therapy by either T-cell depleting polyclonal antibodies such as Anti-Thymocyte Globulins (ATG) or non-depleting anti-interleukine 2 receptor monoclonal antibodies (anti-CD25 moAb: basiliximab or daclizumab) are used to prevent acute rejection, especially in highly sensitized patients. Both induction therapy regimens have a different tolerance profile. Infections and haematological side-effects are more frequently reported in patients receiving ATG. With respect to the efficacy, no comparison exists between both induction therapy regimens in high risk immunological patients as actually defined. Within the last few years, the development of new immunological screening tools, i.e. Luminex assay, had lead to a better evaluation of the immunological status of candidates for kidney transplantation, mainly those who were considered as highly sensitized. The aim of our pilot study is to evaluate ATG and basiliximab induction therapy in de novo sensitized kidney-transplant patients (incompatible grafts rate ≥ 50%) without Donor Specific Antibodies (DSAs) detected by Luminex. Maintenance immunosuppressive regimen will be based on the combination of tacrolimus, mycophenolate sodium and steroids. The primary endpoint is a composite of biopsy-proven acute rejection, graft loss, loss of follow up, or death at 6 months post-transplant. The secondary endpoints are the efficacy of the therapy at month 12 posttransplant, and safety parameters (CMV infection, BK virus nephropathy, haematological tolerance, Adverse Events (AE)and Serious Adverse Events (SAE)). Our hypothesis is that basiliximab induction therapy may be sufficiently effective to prevent acute rejection in sensitized patients without DSA. This may reduce the post-transplant immunosuppression-induced side-effects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged from 18 to 70 years
* Recipient of a deceased or living donor kidney transplant with the following criteria:
* Incompatible grafts rate ≥ 50% for the last available serum before transplantation < 3 months
* Anti-HLA antibodies positive
* Negative DSA by luminex method on historical serum and day serum
* T and B negative Cross match on historical and day serum
* Females capable of becoming pregnant must have a negative serum pregnancy test within 7 days prior to or at screening, and are required to practice an approved and reliable method of birth control for the duration of the study and for a period of 2 months after study medication discontinuation, even where there has been a history of infertility
* Patients who are willing and able to participate in the full course of the study and from whom written informed consent has been obtained.
* Patients affiliated to, or recipients of, a social security system

Exclusion Criteria:

* Recipients of a multi-organ transplantation, including dual kidneys, or who have previously received non renal transplanted organs
* Recipients of a kidney from non-heart beating donor, or with ABO incompatibility against the donor or with a T positive cross match
* Patients with severe uncontrolled systemic infection or severe allergy requiring acute or chronic treatment
* Aspartate aminotransferase (ASAT), Alanine Amino Transferase (ALAT) or bilirubin ≥ 3 upper limit of the normal range (ULN)
* Known hypersensitivity or contra-indication to rabbit proteins, basiliximab, tacrolimus, mycophenolic acid or any of the product excipients
* Patients who are Hepatitis C positive (positive PCR and normal hepatic test may be included), HIV positive, or Hepatitis B surface antigen positive (AgHBs).
* Patients with thrombocytopenia < 75,000/mm3, an absolute neutrophils count < 1,500/mm3, leukocytopenia < 2,500/mm3, and/or hemoglobin < 8g/dL at inclusion visit
* Patients with any past or present malignancy within the last five years except excised squamous or basal cell carcinoma of the skin and treated in situ cervix uteri cancer
* Any surgical or medical condition, excluding transplantation which compromise the inclusion of the patient (investigator's opinion)
* Female patients who are pregnant, breast feeding or capable to become pregnant and not wishing or capable to practice a medically approved and reliable method of birth control
* Patients with symptoms of significant somatic or mental illness. Inability to cooperate or communicate with the investigator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-09; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment failure | 6 months
  Incidence of treatment failure (Biopsy Proved Reject, lost to follow up, graft loss or death) at 6 months post transplantation.

SECONDARY OUTCOMES:
feasibility estimating the number of informed consent obtained | 12 months
  Estimating the number of informed consent obtained
treatment efficacy | 12 months
  Treatment failure at 12 months post transplantation.
  * premature discontinuation of study medication, discontinuation from the study and reasons.
  * incidence of all acute rejection episodes requiring an anti-T and /or anti-B antibodies treatment within 12 months post transplantation.
  * Incidence of C4d positive biopsy findings.
  * Renal function at 3, 6 and 12 months post transplantation (abbreviated MDRD, serum creatinine and adjusted Cockcroft- Gault).
adverse events | 12 months
  Safety:
  - Adverse Events, Serious Adverse Events
patient enrolled in each center | 12 months
  Estimating the number of patient enrolled in each center and by year
number of patients lost from follow-up | 12 months
  Estimating the number of patients lost from from follow-up before 6 and before 12 months
rejection | 12 months
  acute rejection at 6 and 12 months post transplantation
  - Subclinical rejection at the 3 month per protocol renal biopsy.
Donor Specific Antibodies | 12 months
  Donor Specific Antibodies at D0, M3 and M12.
Incidence of BKV viremia | 12 months
  incidence of BKV viremia at 1, 3, 6 and 12 months post transplantation
values of hematologia : hemoglobine, leucocytes, plaquettes, hematies, neutrophiles | 12 months
Incidence of BKV nephropathy | 12 months
  Incidence of BKV nephropathy at 1, 3, 6 and 12 months post transplantation
incidence of CMV post transplantation | 12 months
  incidence of CMV(PCR) post transplantation at 6, 9 and 12 months
incidence of infections | 12 months
  incidence of infections cancer and PTLD

CONTACTS AND LOCATIONS:
Overall Officials: Nassim Kamar, MD PhD, Study Chair — University Hospital, Toulouse
Locations (1):
- UHToulouse, Toulouse, France, France

REFERENCES:
- [Result] Kamar N, Lepage B, Couzi L, Albano L, Durrbach A, Pernin V, Esposito L, Hebral AL, Darres A, Lequintrec M, Cassuto E, Merville P, Congy N, Del Bello A. A Randomized Prospective Study Comparing Anti-T-Lymphocyte Igs to Basiliximab in Highly Sensitized Kidney Transplant Patients. Kidney Int Rep. 2020 Jun 2;5(8):1207-1217. doi: 10.1016/j.ekir.2020.05.020. eCollection 2020 Aug. PMID 32775820